CLINICAL TRIAL: NCT07175662
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of NWRD08 in Patients With HPV16/18-Positive Cervical High-Grade Squamous Intraepithelial Lesion (HSIL)
Brief Title: Evaluation of NWRD08 for HPV-16 and/or HPV-18 Related Cervical HSIL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Newish Biotech (Wuxi) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NWRD08-201
Record Dates: First submitted 2025-09-01; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: High-grade Squamous Intraepithelial Lesion (HSIL)
Keywords: cervical HSIL; NWRD08; HPV16; HPV18
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2mg NWRD08 (Experimental): Each patient will be administered NWRD08 by electroporation at Week0, 4, 8, and 16.
  Interventions: Biological: NWRD08 administered by electroporation
- 4mg NWRD08 (Experimental): Each patient will be administered NWRD08 by electroporation at Week0, 4, 8, and 16.
  Interventions: Biological: NWRD08 administered by electroporation
- Placebo for the 2 mg NWRD08 arm (Placebo Comparator): Each patient will be administered Placebo control by electroporation at Week 0, 4, 8, and 16.
  Interventions: Biological: Placebo administered by electroporation
- Placebo for the 4 mg NWRD08 arm (Placebo Comparator): Each patient will be administered Placebo control by electroporation at Week 0, 4, 8, and 16.
  Interventions: Biological: Placebo administered by electroporation

INTERVENTIONS:
Biological: NWRD08 administered by electroporation — NWRD08 delivered via IM injection + electroporation using TERESA device
  Arms: 2mg NWRD08; 4mg NWRD08
Biological: Placebo administered by electroporation — Placebo delivered via IM injection + electroporation using TERESA device
  Arms: Placebo for the 2 mg NWRD08 arm; Placebo for the 4 mg NWRD08 arm

SUMMARY:
This is a randomized, double-blind, placebo controlled Phase 2 study to determine the efficacy and safety of NWRD08 administered by intramuscular (IM) injection followed by electroporation (EP) in adult women with histologically confirmed cervical high grade squamous intraepithelial lesion (HSIL) (cervical intraepithelial neoplasia grade 2 [CIN2] or grade 3 [CIN3]) associated with human papillomavirus (HPV) 16 and/or HPV18.

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy and safety of NWRD08 in patients with HPV16 and/or HPV18 positive cervical high-grade squamous intraepithelial lesion (HSIL). Eligible subjects will be randomized in a 2:2:1:1 ratio to four arms: 2 mg NWRD08, 4 mg NWRD08, and their respective matching placebo arms.

Participants will receive intramuscular injections of either NWRD08 or matching placebo at the corresponding dose at Week0, 4, 8, and 16 (a total of 4 doses).

Efficacy evaluations at Week 36 will include colposcopy, histopathological biopsy, cervical cytology, and HPV testing.

ELIGIBILITY:
Inclusion Criteria:

Subjects had to meet all of the following inclusion criteria:

1. Aged 18 to 60 years, female.

2. Confirmed by the central laboratory, histopathology results demonstrated cervical HSIL with concurrent HPV16 and/or HPV18 positivity.

3. Colposcopy results during screening must meet the following criteria:

1. The colposcopy must be satisfactory, allowing clear visualization of the entire acetowhite area or the extent of suspected cervical intraepithelial neoplasia (CIN) lesions, including the upper border of the lesion.
2. If the upper border of the lesion is unclear, endocervical curettage (ECC) results must be negative.
3. The cervical lesion area must be less than 75% of the surface of the ectocervix.

4. Fully understand the study and voluntarily sign the informed consent form, able to communicate well with the investigator and complete all treatments, examinations, and visits as required by the study protocol. The informed consent form must be signed before performing any study-specific procedures.

5. At screening, the investigator judges the electrocardiogram (ECG) as normal or without clinically significant findings.

6. Normal function of major organs within 1 week before the first dose: Blood routine: Hemoglobin (Hb) ≥100 g/L; platelet count (PLT) ≥75×10⁹/L; white blood cell count (WBC) ≥3.0×10⁹/L; absolute neutrophil count (ANC) ≥1.5×10⁹/L.

Liver: Total bilirubin (TB) ≤1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 × ULN; plasma albumin ≥30 g/L.

Kidney: Serum creatinine (Scr) ≤1.5 × ULN, or creatinine clearance rate ≥60 mL/min (calculated by Cockcroft-Gault formula) (if serum creatinine >1.5 × ULN).

7. Women of childbearing potential must be willing to consistently and correctly use a contraceptive method with a failure rate of less than 1% per year from the time of signing the informed consent form until the end of the study. Acceptable methods include:

1. Hormonal contraceptives: Combined or progestin-only methods, including oral contraceptives, injections, implants, vaginal rings, or transdermal patches. Subjects with a history of hypercoagulable states (e.g., deep vein thrombosis, pulmonary embolism) must not use hormonal contraceptives.
2. Abstinence from penile-vaginal intercourse.
3. Intrauterine device (IUD) or intrauterine system (IUS).
4. Female subject's male partner sterilized for at least 6 months prior to study entry, and this male is the subject's sole sexual partner.
5. Condom use, with emergency contraception required in case of accidents such as slippage or breakage.
6. Postmenopausal patients (defined as at least 12 consecutive months of amenorrhea without alternative medical causes, with serum follicle-stimulating hormone levels within the laboratory reference range for postmenopausal women) or those sterilized for more than 12 months prior to screening may be considered not requiring contraception.

Exclusion Criteria:

Patients with any of the following were excluded from the study:

1. Any histopathologically confirmed cervical adenocarcinoma/adenocarcinoma in situ (AIS), high-grade vulvar, vaginal, or anal intraepithelial lesions or invasive cancer.
2. Female participants who are pregnant, breastfeeding, or planning to become pregnant during the study.
3. Administration of any live vaccine within 4 weeks prior to the first dose and/or any non-live vaccine within 2 weeks prior to the first dose.
4. Use of blood or blood-related products (including immunoglobulins) within 3 months prior to the first dose or planned use during the study.
5. Prior receipt of therapeutic HPV vaccines (excluding prophylactic HPV vaccines) before screening.
6. Treatment for cervical HSIL within 4 weeks prior to the first dose.
7. Presence of metal implants or implantable medical devices within the electroporation area.
8. Participation in another clinical trial within 30 days prior to screening or being in the follow-up period of another clinical trial.
9. Continuous (for more than 1 week) systemic treatment with corticosteroids (at a dose equivalent to >10 mg/day prednisone or equivalent doses of other corticosteroids) or other immunosuppressive drugs within 30 days prior to screening, with the following exceptions.

   1. Inhaled, ophthalmic, or topical use of corticosteroids at doses ≤10 mg/day prednisone or equivalent is permitted.
   2. Physiological corticosteroid replacement therapy at doses ≤10 mg/day prednisone or equivalent is permitted.
10. History of immunodeficiency or autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, etc.) or current active autoimmune diseases requiring systemic treatment (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressive drugs).
11. Current or anticipated use of disease-modifying antirheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate) and biologic disease-modifying drugs (e.g., infliximab, adalimumab, etanercept) during the study.
12. Continuous (for more than 1 week) use of immunosuppressants such as cyclosporine, tacrolimus, azathioprine, 6-mercaptopurine, and antilymphocyte globulin, as well as other inhibitors affecting immune function (e.g., IL-6 inhibitors, TNF inhibitors, IL-17/23 inhibitors, JAK inhibitors) within 30 days prior to screening.
13. History of solid organ or bone marrow transplantation.
14. Active infections requiring systemic treatment (including active tuberculosis, active Treponema pallidum infection, and bacterial, fungal, or viral infections requiring systemic therapy).
15. Positive test results for any of the following: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), Treponema pallidum antibody (TP-Ab), or human immunodeficiency virus antibody (anti-HIV).
16. Participants with active herpes zoster virus infection.
17. Participants with severe dysfunction of other organs or cardiopulmonary diseases.
18. Epilepsy requiring medication (e.g., steroids or antiepileptic drugs).
19. History or current diagnosis of malignancy.
20. History of severe allergies, allergic diseases, or allergic constitution, meeting any of these criteria.
21. Evidence or history of clinically significant cardiac disease, including but not limited to:

1) Congestive heart failure (NYHA Class >2). 2) Unstable angina. 3) Myocardial infarction within the past 3 months. 4) Any supraventricular or ventricular arrhythmia requiring treatment or intervention.

5) QTc interval ≥470 ms. 6) Poorly controlled hypertension (defined as systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg while on antihypertensive medication).

22. Known psychiatric or substance abuse disorders that may interfere with the subject's ability to comply with study requirements.

23. History or current evidence of any condition, treatment, laboratory abnormality, or other circumstance that may increase the risk associated with study participation or study intervention administration, or may interfere with the interpretation of study results, and which, in the investigator's judgment, makes the subject unsuitable for enrollment in this study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Histopathological Regression of Cervical Lesions to CIN 1 or no lesions at week 36 | Week 36
  The number of participants with histopathologically confirmed CIN2/3 or CIN 3 associated with HPV16 or HPV18 whose cervical lesions regress to CIN 1 or no lesions at the 36 week visit.

SECONDARY OUTCOMES:
Incidence and severity of local and systemic adverse events (AEs). | up to 40 weeks
  Adverse events (AEs) and serious adverse events (SAEs) will be monitored based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Incidence and severity of adverse events (AEs) at the injection site. | up to 40 weeks
  Adverse events (AEs) and serious adverse events (SAEs) will be monitored based on the Guidance on Grading Standards for Adverse Events in Clinical Trials of Preventive Vaccines.
Incidence and severity of all serious adverse events (SAEs). | up to 40 weeks
  Incidence and severity of all serious adverse events (SAEs) during the study period (e.g., suspected unexpected serious adverse reactions, unexpected adverse device effects).
Pregnancy occurrences and outcomes during the study period | up to 40 weeks
Incidence of investigational product-related adverse events (AEs) leading to treatment discontinuation. | up to 40 weeks
Incidence of Grade 3 or higher adverse events (AEs) related to the investigational product. | up to 40 weeks
Proportion of Participants with Histopathological Regression to no lesions. | Week 36
  The number of participants with histopathologically confirmed CIN2/3 or CIN 3 associated with HPV16 or HPV18 whose cervical lesions regress to no lesions at the 36 week visit.
Proportion of Participants with Histopathological Regression to LSIL/CIN1. | Week 36
  The number of participants with histopathologically confirmed CIN2/3 or CIN 3 associated with HPV16 or HPV18 whose cervical lesions regress to LSIL/CIN1 at the 36 week visit.
Proportion of Participants with Virologically-proven Clearance of HPV 16 and/or HPV18. | Week 36
  The number of participants with virologically-proven clearance of HPV16 and/or HPV18 at the 36 week visit.
Proportion of Participants with Virologically-proven Clearance of HPV 16 or HPV18 or Histopathological Regression of Cervical Lesions to LSIL/CIN 1 or no lesion. | Week 36
  The number of participants with Virologically-proven Clearance of HPV 16 or HPV18 or Histopathological Regression of Cervical Lesions to LSIL/CIN 1 or no lesion at the 36 week visit.
Proportion of Participants with Virologically-proven Clearance of HPV 16 or HPV18 in Combination with Histopathological Regression of Cervical Lesions to LSIL/CIN 1 or no lesion. | Week 36
  The number of participants with Virologically-proven Clearance of HPV 16 or HPV18 in Combination with Histopathological Regression of Cervical Lesions to LSIL/CIN 1 or no lesion at the 36 week visit.
Proportion of Participants with Virologically-proven Clearance of HPV 16 or HPV18 in Combination with Histopathological Regression of Cervical Lesions to no lesion. | Week 36
  The number of participants with Virologically-proven Clearance of HPV 16 or HPV18 in Combination with Histopathological Regression of Cervical Lesions to no lesion at the 36 week visit.
Levels of cellular immune responses. | Week 10, 18, 24, and 36
  Levels of cellular immune responses measured by interferon-gamma enzyme-linked immunospot (IFN-γ ELISPOT) assay in peripheral blood mononuclear cells (PBMCs) of subjects at baseline and at Week 10, 18, 24, and 36 after first dose.
Levels of serum anti-HPV16 and anti-HPV18 antibody titers. | Week 10, 18, 24, and 36
  Levels of serum anti-HPV16 and anti-HPV18 antibody titers measured in peripheral blood samples collected at baseline and at Week 10, 18, 24, and 36 after initial vaccination.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Institute and Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided